CLINICAL TRIAL: NCT05228548
Title: Development and Interpretation of a Machine Learning Model for Perioperative Transfusion Prediction
Brief Title: Machine Learning Model for Perioperative Transfusion Prediction
Status: Completed | Type: Observational
Sponsor: Diskapi Teaching and Research Hospital (Other)
Collaborators: Hacettepe University (Other); Dokuz Eylul University (Other); Saglik Bilimleri Universitesi (Other); Bulent Ecevit University (Other); Erzincan University (Other); Kahramanmaras Sutcu Imam University (Other); Ufuk University (Other); Istanbul Medeniyet University (Other); Marmara University (Other); Eskisehir Osmangazi University (Other); Inonu University (Other); Mersin University (Other); Istanbul University (Other); Selcuk University (Other); Balikesir University (Other); Trakya University (Other); Necmettin Erbakan University (Other); Ankara University (Other); Suleyman Demirel University (Other); Tobb University of Economics and Technology (Other); Akdeniz University (Other); Uludag University (Other); Ordu University (Other); Gazi University (Other); TC Erciyes University (Other); Hitit University (Other); Firat University (Other); Karadeniz Technical University (Other); Ondokuz Mayıs University (Other); Yuzuncu Yil University (Other); Namik Kemal University (Other); Baskent University (Other); Celal Bayar University (Other); Osmaniye Government Hospital (Other Government)
Responsible Party: Principal Investigator, DILEK YAZICIOGLU, Prof. Dr. Dilek Unal, Diskapi Teaching and Research Hospital
Other Study IDs: Machine learning DiskapiTRH
Record Dates: First submitted 2022-01-13; First posted 2022-02-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-01

CONDITIONS: Surgery; Blood Transfusion
Keywords: Decision tree; eXtreme garadient boosting; k-nearest neighbors; Logistic regression; Machine learning; Prediction model; Random forest; Red blood cell transfusion; Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Perioperative blood transfusion — Perioperative blood transfusion

SUMMARY:
This study aimed to develop and interpret a machine learning model to predict red blood cell (RBC) transfusion.

DETAILED DESCRIPTION:
A dataset from a multicenter study involving 6121 patients underwent elective major surgery was analysed. Data concerning patients who received inappropriate RBC transfusion were excluded. Twenty one perioperative features were used to predict RBC transfusion. The data set was randomly split into train and validation sets (70-30). Decision tree, random forest, k-nearest neighbors, logistic regression, and eXtreme garadient boosting (XGBoost) methods were used for prediction. The area under the curves (AUC) of the receiver operating characteristics curves for the machine learning models used for RBC transfusion prediction were compared.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Underwent major elective surgery

Exclusion Criteria:

* Pediatric patients
* Emergency cases

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing major elective surgical procedures were considered eligible. All age groups and both genders were included. The surgical procedures were predefined according to the Classification of Diagnostic, Therapeutic, and Surgical Procedures of the National Social Insurance Institution, in which every procedure has a unique cod
Sampling Method: Non-Probability Sample
Enrollment: 6121 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Number of patients received Red blood cell transfusion | Perioperative period
  Number of patients received Red blood cell transfusion
The area under the curve | Perioperative period
  The the area under the curve of the receiver operating characteristics curves

CONTACTS AND LOCATIONS:
Overall Officials: Dilek D Unal, Prof, Principal Investigator — UNIVERSITY OF HEALTH SCIENCES TURKEY DISKAPI YILDIRIM BEYAZIT TRAINING RESEARCH HOSPITAL ANKARA
Locations (1):
- Dilek D Unal, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Murphy GJ, Reeves BC, Rogers CA, Rizvi SI, Culliford L, Angelini GD. Increased mortality, postoperative morbidity, and cost after red blood cell transfusion in patients having cardiac surgery. Circulation. 2007 Nov 27;116(22):2544-52. doi: 10.1161/CIRCULATIONAHA.107.698977. Epub 2007 Nov 12. PMID 17998460
- [Result] Bernard AC, Davenport DL, Chang PK, Vaughan TB, Zwischenberger JB. Intraoperative transfusion of 1 U to 2 U packed red blood cells is associated with increased 30-day mortality, surgical-site infection, pneumonia, and sepsis in general surgery patients. J Am Coll Surg. 2009 May;208(5):931-7, 937.e1-2; discussion 938-9. doi: 10.1016/j.jamcollsurg.2008.11.019. Epub 2009 Mar 26. PMID 19476865
- [Result] Walczak S, Velanovich V. Prediction of perioperative transfusions using an artificial neural network. PLoS One. 2020 Feb 24;15(2):e0229450. doi: 10.1371/journal.pone.0229450. eCollection 2020. PMID 32092108